CLINICAL TRIAL: NCT05645510
Title: LIVInG With chrONic Cancer TrEatments (LONGEVITI) Study
Acronym: LONGEVITI
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC-22-0196
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Tyrosine Kinase Mutation; Breast Cancer; Melanoma; Multiple Myeloma; Chronic Leukemia; Prostate Cancer; Ovarian Cancer; Colorectal Cancer; Lung Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Melanoma; Multiple Myeloma; Prostatic Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with advanced chronic cancers are now living for many years as a result of new targeted anti-cancer treatments. Many of these treatments are quite new and people may take them for months, even years, as long as the treatments are helping. The purpose of this study is to help understand how to best support people receiving these treatments.

DETAILED DESCRIPTION:
Participants ill be scheduled for an in-person, telephone or computer video interview with the researcher(s). They will be asked about their experiences receiving targeted anti-cancer treatments. Then over the next 3 months, participants will be asked to think about how receiving these cancer treatments affects daily living and to create a 'metaphor'. Metaphors may be composed with any mix of visual, verbal, musical or other works participants feel expresses and brings their experiences to life.

ELIGIBILITY:
Inclusion Criteria: taking chronic targeted anti-cancer agents -

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with cancer taking oral anti-cancer agents over the long term
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Interview | 3 months
  Interview to learn the experiences of people living with incurable cancers

CONTACTS AND LOCATIONS:
Locations (1):
- Edith Pituskin, Edmonton, Alberta, Canada